CLINICAL TRIAL: NCT05513664
Title: To Evaluate Real-World Effectiveness of Osimertinib for Patients With Advanced or Metastatic Epidermal Growth Factor Receptor 20exon Insertion Mutation (20ins) Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Real-World Effectiveness of Osimertinib for Patients With Non-Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Collaborators: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: JMT101-010
Record Dates: First submitted 2022-08-23; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-07

CONDITIONS: Locally Advanced or Metastatic Non-Small Cell Lung Cancer; EGFR Exon20 Insertion Mutations
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Osimertinib — 80 or 160 mg/qd

SUMMARY:
This study is a retrospective real-world study to evaluate the efficacy of Osimertinib for patients with advanced or metastatic EGFR 20exon insertion mutation (20ins) Non-Small Cell Lung Cancer.

DETAILED DESCRIPTION:
This is a multicenter, retrospective observational real-world study, which evaluates the efficacy of Osimertinib, between 2017 and 2022, in patients with advanced or metastatic EGFR 20exon insertion mutation (20ins) Non-Small Cell Lung Cancer. This study serves as the external control for a single arm phase II trial on JMT101 combined with Osimertinib in patients with Non-Small Cell Lung Cancer. The primary outcome measure is objective response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced or metastatic (stage ШB-Ⅳ, 8th AJCC) NSCLC confirmed by histology or cytology;
2. The result of EGFR 20ins is positive detected by tissue, blood, pleural fluid or cerebrospinal fluid;
3. Have received osimertinib treatment after detection of EGFR 20ins;
4. Age of 18 years or above;
5. Information about tumor outcome evaluation is required at least once after osimertinib treatment (such as tumor imaging data, description of efficacy evaluation in medical records, etc.).

Exclusion Criteria:

1. Previously treated with JMT101 (Patients will be included if osimertinib treatment is before JMT101 treatment);
2. Patients harboring EGFR exon20 insertion mutation and also have other EGFR TKI-sensitizing EGFR mutations, such as G719X mutation in exon 18, exon 19 deletion mutation (19 del), exon 20 T790M or S768I mutation, exon 21 L858R mutation, or L861Q mutation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received osimertinib with advanced or metastatic EGFR 20exon insertion mutation (20ins) Non-Small Cell Lung Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
1.Real world Objective Response Rate (rwORR) | March 2017 to May 2022

SECONDARY OUTCOMES:
Real world Duration of Response（rwDOR） | From March 2017 to May 2022
Real world Disease Control Rate（rwDCR） | From March 2017 to May 2022
Real world Progression Free Survival（rwPFS） | From March 2017 to May 2022

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - Affiliated Hospital of Hebei University, Baoding
  - Beijing Cancer Hospital, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Chinese People's Liberation Army General Hospital, Beijing
  - Chongqing Cancer Hospital, Chongqing
  - Southwest Hospital of Army Medical University, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - Anhui Cancer Hospital, Hefei
  - Shandong Cancer Hospital, Jinan
  - Nanjing Chest Hospital, Nanjing
  - Fudan University Cancer Hospital, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Shanxi Provincial People's Hospital, Shanxi
  - The Fourth Hospital of Hebei Medical University, Shijia Zhuang
  - West China Hospital of Sichuan University, Sichuan
  - Shanxi Cancer Hospital, Taiyuan
  - Huazhong University of Science Tongji Hospital, Tongji Medical College, Wuhan
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Henan Cancer Hospital, Zhengzhou